CLINICAL TRIAL: NCT00054912
Title: An Open Label, Multi-Center Safety and Tolerance Study of EP2101 Peptide Vaccine in Patients With Stage III Colon Cancer
Brief Title: An Open Label Study of a Peptide Vaccine in Patients With Stage III Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epimmune (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP2101-102
Record Dates: First submitted 2003-02-12; First posted 2003-02-14 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2004-04

CONDITIONS: Colonic Neoplasms; Colorectal Neoplasms
Keywords: vaccine; colon; cancer; colorectal; neoplasm; Colonic Cancer; Colon Cancer; Cancer of the Colon
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Neoplasms

INTERVENTIONS:
Biological: EP2101

SUMMARY:
EP2101 is a new cancer vaccine containing 10 different peptide antigens. The vaccine is designed to activate the immune system to develop a response against tumor cells in order to delay or prevent the recurrence of cancer. This study will test the safety and measure the level of immune stimulating capability of EP2101 in patients with Colon Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Colon Cancer, stage III
* At least four weeks following prior standard treatment, with no evidence of disease
* Must use adequate birth control

Exclusion Criteria:

* Prior cancer vaccine therapy or concurrent participation in any other investigational study
* A history of HIV, Hepatitis B or C, or any other acute medical condition which may compromise patient safety or the activity of the study vaccine treatment
* A history of adverse reactions following administration of any vaccines, or a history of hypersensitivity to any components of the study vaccine
* Women who are pregnant, intend to become pregnant, or who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-02

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Southern California School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Cancer Centers of Florida, Orlando, Florida
  - New York Oncology Hematology, Albany, New York
  - Duke University Medical Center, Durham, North Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - University of Washington, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.idm-biotech.com